CLINICAL TRIAL: NCT02060357
Title: Comparison of Two New Generation Drug Eluting Stents in Patients With Diabetes
Brief Title: Comparison of Two New Generation Drug Eluting Stents in Patients With Diabetes (OCT-DES)
Acronym: OCT-DES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Barts & The London NHS Trust (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Principal Investigator, Anthony Mathur, Professor, Barts & The London NHS Trust
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: 11/LO/0948
Record Dates: First submitted 2014-01-20; First posted 2014-02-12 (Estimated); Last update posted 2015-08-07 (Estimated); Status verified 2015-08

CONDITIONS: Coronary Artery Disease; Diabetes
Keywords: Diabetes Mellitus; PCI; Drug eluting stent; OCT
MeSH Terms: conditions — Coronary Artery Disease; Diabetes Mellitus | interventions — Tomography, Optical Coherence

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Resolute Integrity Stent (Active Comparator): Patients will be randomised in a 1:1 ratio to receive two different types of DES
  Interventions: Device: Optical coherence tomography
- Promus Stent (Active Comparator): Patients will be randomised in a 1:1 ratio to receive two different types of DES
  Interventions: Device: Optical coherence tomography

INTERVENTIONS:
Device: Optical coherence tomography

SUMMARY:
The aim of this study is a comparative evaluation of re-endothelailisation of the Integrity Resolute zotarolimus eluting stent (Medtronic) and of the Promus Element erolimus eluting stent (Boston Scientific), in patients with diabetes.

We plan to compare endothelial coverage and neointimal proliferation using OCT and compare this data to published results from conventional stents.

ELIGIBILITY:
Inclusion Criteria:

* Known to have diabetes
* Scheduled for percutaneous coronary intervention (PCI) with a stenosis suitable for DES implantation and OCT imaging
* Reference vessel diameter over 2.5mm by operator assessment.
* Able to understand and sign the written Informed Consent Form.
* Able and willing to follow the Protocol requirements.

Exclusion Criteria:

* Inability to consent
* Cardiogenic shock
* Planned use of a bare metal stent
* LMS coronary artery disease
* Congestive cardiac failure or low ejection fraction (LVEF <35%)
* Lesions unsuitable for OCT
* Total length of stented lesion greater than 55mm (total combination of stent lengths)
* Age less than 18 years or age greater than 80 years
* Planned surgical procedure ≤ 12 months post PCI procedure
* Patient demonstrates evidence of thrombocytopenia (platelet count < 100,000/mm3)
* Patients with contraindications to ASA, clopidogrel, or prasogrel
* Patient is currently on warfarin, or possibility of treatment with warfarin during the following 12 months post index procedure
* Allergy to contrast
* Patients enrolled in another active clinical trial.
* Potential for non-compliance towards the requirements in the study protocol.
* Serious known concomitant disease with a life expectancy of less than one year
* Follow-up impossible (no fixed abode, etc)
* Patients with renal impairment (Creatinine >200mmol/L)
* Subjects of childbearing potential

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-11; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Endothelial stent coverage | 6 month
  Endothelial coverage expressed as % of struts without coverage as measured by OCT

SECONDARY OUTCOMES:
Neointimal hyperplasia | 6 month
  Neointimal hyperplasia (mm2) as measured by OCT
MACE | 6 months
  death, heart failure, myocardial infarction, stroke, need for repeat revascularisation

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Mathur, FRCP FESC, Principal Investigator — Barts & The London NHS Trust
Locations (1):
- London Chest Hospital, Barts Health NHS Trust, London, United Kingdom

REFERENCES:
- [Derived] Hamshere S, Byrne A, Choudhury T, Gallagher SM, Rathod KS, Lungley J, Knight CJ, Kapur A, Jones DA, Mathur A. Randomised trial of the comparison of drug-eluting stents in patients with diabetes: OCT DES trial. Open Heart. 2018 Apr 5;5(1):e000705. doi: 10.1136/openhrt-2017-000705. eCollection 2018. PMID 29632674